CLINICAL TRIAL: NCT06466577
Title: Clinical Study of CT 5400 RT for System Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Philips Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200254
Record Dates: First submitted 2024-04-09; First posted 2024-06-20 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Performance and Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Image quality performance (Other)
  Interventions: Diagnostic Test: CT 5400 RT System

INTERVENTIONS:
Diagnostic Test: CT 5400 RT System — Computed Tomography X-RAY System is intended to produce images of the head and body by computer reconstruction of x-ray transmission data taken at different angles and planes.

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of the CT 5400 RT System.

ELIGIBILITY:
Inclusion Criteria:

* 18≤ Age ≤ 75 years old;
* Subjects with Clear consciousness; Subjects can cooperate and act autonomously;
* Subjects agree to participate in this clinical study and sign the subject's informed consent;
* Women subjects of childbearing age should have a negative pregnancy test and should have no plans to become pregnant in the next 6 months.

Exclusion Criteria:

* Subjects who do not have full capacity for civil conduct;
* Women subjects who are pregnant or in lactating phase;
* Subjects who have had a CT scan within one year;
* Subjects with a history of allergies or asthma, severe hepatic and renal insufficiency or hyperthyroidism in which are considered as contraindication for CT contrast-enhanced examination;
* According to the opinion of the investigator: any situation that may affect the evaluation of the results or expose subjects into health risk;
* Subjects with mental disorders who cannot cooperate with the examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Clinical image quality | 14 days (anticipated)
  Image quality will be assessed by Likert score (1-5)

SECONDARY OUTCOMES:
General function assessment | 14 days (anticipated)
  A three-scale assessment will be used for Image exposure level, couch movement, speaker& microphone voice quality, image post processing capability, data storage.
  A three-scale criteria- Very satisfied, Satisfied, Dissatisfied
  Assessment criteria: all parameters will be assessed based on the user's feelings. The parameters should all reach "Satisfied", indicating that the general function of the case meet the clinical application requirements.
Convenience assessment | 14 days (anticipated)
  A three-scale assessment will be used for laser positioning, panel control, user-friendly interface of post-processing software, operation of post-processing software.
  A three-scale criteria- Very satisfied, Satisfied, Dissatisfied
  Assessment criteria: all parameters will be assessed based on the user's feelings. The parameters should all reach "Satisfied", indicating that the general function of the case meet the clinical application requirements.
Workflow and stability assessment | 14 days (anticipated)
  A three-scale assessment will be used for workflow, Image display and transmission, system inactivation, unexpected system shutdown, unexpected termination during scanning, fail to expose during scanning
  A three-scale criteria- Very satisfied, Satisfied, Dissatisfied
  Assessment criteria: all parameters will be assessed based on the user's feelings. The parameters should all reach "Satisfied", indicating that the general function of the case meet the clinical application requirements.
Incidence of CT Scan-Emergent Adverse Events | 30 days (anticipated)
  Monitor adverse events and serious adverse events(safety and tolerance) during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No